CLINICAL TRIAL: NCT07176780
Title: Effect of Semiconductor Embedded Wearable Sleeve on the Treatment and Mitigation of Primary Dysmenorrhea Symptoms: A Randomized, Double-Blinded, Placebo-Controlled Clinical Trial
Brief Title: Effect of Semiconductor Embedded Wearable Sleeve on Treatment of Primary Dysmenorrhea Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: INCREDIWEAR HOLDINGS, INC. (Industry)
Responsible Party: Principal Investigator, Anne Flynn, MD, Assistant Clinical Professor, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2264207
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Primary Dysmenorrhea; Primary Dysmenorrhea (PD); Menstrual Cramps; Women's Health
Keywords: Menstrual Cramps; Dysmenorrhea; Primary Dysmenorrhea; Women's Health
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Device (Active Comparator): Device embedded with semiconductors
  Interventions: Device: Semiconductor embedded body sleeve
- Placebo Device (Placebo Comparator): Identical device absent of semiconductors
  Interventions: Device: Placebo Non-Compressive Body Sleeve

INTERVENTIONS:
Device: Semiconductor embedded body sleeve — The active device contains semiconductors embedded into the body sleeve fabric
  Arms: Active Device
Device: Placebo Non-Compressive Body Sleeve — Identical body sleeve absent of semiconductors
  Arms: Placebo Device

SUMMARY:
This study is looking to test a non-compressive semiconductor embedded body sleeve for treatment of primary dysmenorrhea symptoms. Dysmenorrhea is the lower abdominal pain (sometimes referred to as "cramping") experienced during menstruation (monthly "period"), affecting up to 94% of people aged from 10-20 years old. The semiconductor embedded fabric increases blood circulation through activation of the embedded elements with body heat while worn and releases energy waves as well as negative ions. This energy has an effect inside the body that increases oxygen and nutrient flow to tissues, and can help to decrease pain and inflammation. This study is testing this technology to see if it can be used as a non-pharmacological treatment for menstrual cramping.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported primary dysmenorrhea during past three menstrual cycles
* Age 18-45 inclusive at the time of consent
* Self-reported typical primary dysmenorrhea symptom pain greater than 4 on a 1-10 visual analog scale (VAS)
* History of regular menstrual cycles with a usual length of 21 to 35 days
* Willing and able to provide informed consent and adhere to study requirements

Exclusion Criteria:

* History of neurological conditions, including multiple sclerosis or Parkinson's disease
* Secondary dysmenorrhea including confirmed or suspected endometriosis or fibroids or intrauterine device
* Self-reported size not available in study device
* Pregnant or planning to become pregnant during the study
* Have within the past six months of enrollment, or are planning to in the next six months, start or discontinue any of the following contraceptive methods:

  1. intrauterine device
  2. oral contraceptives,
  3. contraceptive patch,
  4. implant (Nexplanon),
  5. shot (Depo-Provera),
  6. vaginal ring
* Chronic pain conditions unrelated to primary dysmenorrhea
* Auto-immune or auto-inflammatory diseases
* Has used within the last 90 days or is planning to use nicotine-containing products
* History of metabolic disorders
* Active infection (local or systemic) that, in the opinion of the investigator, would prevent usage of the device
* In the opinion of the investigator, any other criteria or condition that could increase the risk associated with study participation or study treatment or could interfere with the interpretation of study results
* Have taken any investigational drug or used any investigational device within the 30 days prior to consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Participant-Reported Changes in Pain | 6 months
  Reduction in menstrual symptom severity as determined by the Visual Analog Scale (VAS) compared to placebo group:
  Visual Analog Scale for Pain (VAS) Minimum value: 0 (no pain) Maximum value: 10 (worst possible pain)

SECONDARY OUTCOMES:
Participant-Reported Changes in Quality of Life | 6 months
  Improvement in health-related quality of life as determined by the Short Form quality of life enjoyment and satisfaction questionnaire (Q-LES-Q-SF) compared to placebo group.
  Q-LES-Q-SF:
  Lowest score: 14 (indicating very poor quality of life) Highest score: 70 (indicating very good quality of life)
Changes in oral medication intake compared to placebo group | 6 months
  As measured by collecting concomitant medication information at baseline and changes throughout participation in the study.
Changes in Participant Pain Score (SF-MPQ-2) | 6 months
  Changes in participant menstrual pain as determined by menstrual pain questionnaire, Short Form McGill Pain Questionnaire (SF-MPQ-2), compared to placebo group.
  SF-MPQ-2:
  Lowest score: 0 (no pain) Highest score: 10 (worst possible pain)
Changes in participant function in daily life | 6 months
  Changes in participant function/distress as determined by Menstrual Distress Questionnaire (MEDI-Q), compared to placebo group.
  MEDI-Q:
  Lowest score: 0 (no distress) Highest score: 5 (very much distress)
Changes in menstrual symptom duration | 6 months
  Changes in menstrual symptom duration compared to placebo group as reported by participants at each menstrual cycle.